CLINICAL TRIAL: NCT02923414
Title: The Efficiency and Safety of a High Energy Shock Protocol (360-360-360 J) Versus a Standard Escalating Energy Shock Protocol (125-150-200 J) in Cardioverting Atrial Fibrillation
Brief Title: Comparison of High Versus Escalating Shocks in Cardioverting Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Randers Regional Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52187
Record Dates: First submitted 2016-10-03; First posted 2016-10-04 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2018-04

CONDITIONS: Atrial Fibrillation
Keywords: Cardioversion
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard escalating shocks (Active Comparator): Patients will be randomized to a standard escalating shock protocol using the energy settings: 125, 150, 200 J. All cardioversion attempts will be performed using LIFEPAK 20, Physio-Control Inc., Redmond, WA, USA
  Interventions: Device: Standard escalating shocks
- High energy shocks (Active Comparator): Patients will be randomized to a high energy shock protocol using the energy settings: 360, 360, 360 J. All cardioversion attempts will be performed using LIFEPAK 20, Physio-Control Inc., Redmond, WA, USA
  Interventions: Device: High energy shock protocol

INTERVENTIONS:
Device: Standard escalating shocks — 125 J, 150 J, 200 J
  Other Names: LIFEPAK 20, Physio-Control Inc., Redmond, WA, USA
  Arms: Standard escalating shocks
Device: High energy shock protocol — 360 J, 360 J, 360 J.
  Other Names: LIFEPAK 20, Physio-Control Inc., Redmond, WA, USA
  Arms: High energy shocks

SUMMARY:
Atrial fibrillation is the most common heart rhythm disorder. For patients suffering atrial fibrillation direct current cardioversion is performed to reduce patients symptoms and prevent disease progression. The optimal energy selection for biphasic cardioversion is unknown.

We aim to investigate the efficiency and safety of a high energy shock protocol (360 J) versus a standard escalating shock protocol (125-150-200 J) in cardioversion of atrial fibrillation.

DETAILED DESCRIPTION:
The optimal energy selection for biphasic direct current (DC) cardioversion of atrial fibrillation is unknown. The energy delivered should be sufficient to achieve prompt cardioversion but without the risk of inducing any potential injury e.g. skin burns, myocardial stunning or post-cardioversion arrhythmias. The use of an escalating protocol, with a low energy initial shock, has been considered conventional practice, originally to avoid post cardioversion arrhythmias when using monophasic shocks.(1) This practice has been directly transferred to biphasic cardioversion. The European Society of Cardiology 2016 guidelines (2) and the American Heart Association/American College of Cardiology 2014 guidelines on the management of atrial fibrillation (3) do not recommend any specific energy settings, whereas the European Resuscitation Council 2010 guidelines for cardiopulmonary resuscitation (4) recommend a starting energy level of 120-200 J with subsequent escalating energy setting.

Previously, a non-escalating protocol (200 J) (5) has been found to have a significantly higher first shock success resulting in fewer shock deliveries without compromising safety compared with a low energy escalating shock protocol (100-150-200 J). Further, a study found fewer arrhythmic complications with increasing energy suggesting an 'upper limit of vulnerability'. It is well-established that biphasic shocks induce fewer post-shock arrhythmias (6), skin burns (7) and shorter periods of myocardial stunning compared with monophasic shocks.(8) Importantly, no correlation between increasing biphasic energy delivery and any complications was found in these studies. Nonetheless, the efficiency and safety of a high energy shock (360 J) biphasic protocol compared with a conventional low energy escalating protocol is unknown. Accordingly, this study aims to compare the efficiency and safety of a high energy protocol (360-360-360 J) versus a standard escalating protocol (125-150-200 J). We hypothesise that a high energy cardioversion protocol is more effective compared to standard escalating energy protocol, without compromising safety.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age, scheduled for cardioversion of atrial fibrillation. Patients with atrial fibrillation for ≤48 hours may be cardioverted immediately. Patients with atrial fibrillation for >48 hours will be required to have a documented weekly international normalized ratio (INR) ≥2.0 (including within 48 hours of cardioversion) or treatment with non-vitamin K oral anticoagulant for three weeks or longer. Alternatively, a transoesophageal echocardiogram documenting absence of intracardiac thrombi is accepted and cardioversion can be performed on treatment with low molecular weight heparin.

Exclusion Criteria:

* Pregnancy, haemodynamically unstable atrial fibrillation, other arrhythmias than atrial fibrillation, untreated hyperthyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Efficacy: Successful cardioversion | One minute following cardioversion
  Successful cardioversion is defined as the proportion of patients in sinus rhythm one minute after cardioversion or cardioversion attempt (to a maximum of the 3 shocks in the protocol).

SECONDARY OUTCOMES:
Efficacy: First shock success | Following first cardioversion attempt
  Successful cardioversion following the first cardioversion attempt (125 J versus 360 J).
Safety: Arrhythmic events and ECG-changes following cardioversion | Within four hours following cardioversion (until discharge)
  Any post-cardioversion arrhythmias will be recorded using ECG-holtering four hours post cardioversion. Further ECG changes will be measured (sinus node dysfunction, atrioventricular delay, ventricular tachyarrhythmia or ventricular premature complexes, ST-segment deviations and recurrence of AF).
Safety: Skin-discomfort, skin burns or itching | Two hours after cardioversion
  Patients self-assessment of skin discomfort and objective measurement of skin burns or itching.
Safety: Troponin I level changes following cardioversion | Four hours after cardioversion
  To evaluate changes in high sensitive cardiac troponin I levels between a baseline measurement before cardioversion and the level four hours following cardioversion.
Safety: Echocardiographic evaluation following cardioversion | Two hours after cardioversion
  Comparing a baseline echocardiographic evaluation with an evaluation performed two after cardioversion, e.g. left ventricular function using standard echocardiographic measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Løfgren, MD, PhD, Study Director — Randers Regional Hospital; Anders S Schmidt, MB, Principal Investigator — Randers Regional Hospital
Locations (1):
- Randers Regional Hospital, Randers, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lown B. Electrical reversion of cardiac arrhythmias. Br Heart J. 1967 Jul;29(4):469-89. doi: 10.1136/hrt.29.4.469. No abstract available. PMID 6029120
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; ACC/AHA Task Force Members. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines and the Heart Rhythm Society. Circulation. 2014 Dec 2;130(23):e199-267. doi: 10.1161/CIR.0000000000000041. Epub 2014 Mar 28. No abstract available. PMID 24682347
- [Background] Deakin CD, Nolan JP, Sunde K, Koster RW. European Resuscitation Council Guidelines for Resuscitation 2010 Section 3. Electrical therapies: automated external defibrillators, defibrillation, cardioversion and pacing. Resuscitation. 2010 Oct;81(10):1293-304. doi: 10.1016/j.resuscitation.2010.08.008. No abstract available. PMID 20956050
- [Background] Glover BM, Walsh SJ, McCann CJ, Moore MJ, Manoharan G, Dalzell GW, McAllister A, McClements B, McEneaney DJ, Trouton TG, Mathew TP, Adgey AA. Biphasic energy selection for transthoracic cardioversion of atrial fibrillation. The BEST AF Trial. Heart. 2008 Jul;94(7):884-7. doi: 10.1136/hrt.2007.120782. Epub 2007 Jun 25. PMID 17591649
- [Background] Ambler JJ, Deakin CD. A randomized controlled trial of efficacy and ST change following use of the Welch-Allyn MRL PIC biphasic waveform versus damped sine monophasic waveform for external DC cardioversion. Resuscitation. 2006 Nov;71(2):146-51. doi: 10.1016/j.resuscitation.2006.03.017. Epub 2006 Sep 20. PMID 16987583
- [Background] Page RL, Kerber RE, Russell JK, Trouton T, Waktare J, Gallik D, Olgin JE, Ricard P, Dalzell GW, Reddy R, Lazzara R, Lee K, Carlson M, Halperin B, Bardy GH; BiCard Investigators. Biphasic versus monophasic shock waveform for conversion of atrial fibrillation: the results of an international randomized, double-blind multicenter trial. J Am Coll Cardiol. 2002 Jun 19;39(12):1956-63. doi: 10.1016/s0735-1097(02)01898-3. PMID 12084594
- [Background] Deakin CD, Ambler JJ. Post-shock myocardial stunning: a prospective randomised double-blind comparison of monophasic and biphasic waveforms. Resuscitation. 2006 Mar;68(3):329-33. doi: 10.1016/j.resuscitation.2005.07.021. Epub 2005 Dec 27. PMID 16378672